CLINICAL TRIAL: NCT00694564
Title: A Pilot Open-labeled Trial of S-adenosyl Methionine (SAM-e) for Recurrent Abdominal Pain in Children
Brief Title: Evaluation of S-adenosyl Methionine (SAM-e) for Recurrent Abdominal Pain in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huang, Jeannie, M.D. (Individual)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCSD060705; IND 75,404
Record Dates: First submitted 2008-06-06; First posted 2008-06-10 (Estimated); Results first posted 2013-09-13 (Estimated); Last update posted 2018-03-16 (Actual); Status verified 2016-01

CONDITIONS: Abdominal Pain
Keywords: abdominal pain; children
MeSH Terms: conditions — Abdominal Pain | interventions — S-Adenosylmethionine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): This an open-labeled study. All participants will be part of the treatment group and receive SAM-e. S-adenosyl methionine will be dosed as 200 mg tablets with doses ranging from 200 to 1400 mg daily.
  Interventions: Drug: S-adenosyl methionine

INTERVENTIONS:
Drug: S-adenosyl methionine — S-adenosyl methionine will be dosed as 200 mg tablets with doses ranging from 200 to 1400 mg daily.
  Other Names: SAM-e; Mood Plus

SUMMARY:
This pilot study will investigate the efficacy of SAM-e for the treatment of recurrent abdominal pain in children. This will be an open-labeled study and all participants will receive SAM-e therapy. Given that SAM-e has been demonstrated to improve symptoms of depression and pain with minimal side effects as compared to other antidepressant therapy, we hypothesize that SAM-e will reduce pain symptoms among children with recurrent abdominal pain.

ELIGIBILITY:
Inclusion Criteria:

* 8 to 22 years old
* Diagnosed with RAP as verified by a physician, and having at least twice weekly episodes of abdominal pain which cause the patient to withdraw from normal activities.
* At least one month trial on a high fiber diet without resolution of abdominal pain.
* Ambulatory

Exclusion Criteria:

* Focal abdominal pain by history or physical exam, unless a negative (including endoscopic) evaluation has been performed
* Current diagnosis of inflammatory bowel disease, pancreatitis (acute or recurrent), peptic ulcer disease, gastrointestinal infection (unresolved), or ongoing gastrointestinal inflammation.
* Current or recent (within the past year) pregnancy and/or current breastfeeding.
* Current diagnosis of nephropathy or genitourinary disease.
* Blood in stools or emesis (EXCEPTION: blood in the stool secondary to hemorrhoids is not an exclusion criterion).
* Unintentional loss of over 10% body weight over the past 3 months or weight < 100% ideal body weight.
* Recurrent fevers (T>100F) at least once a week or with abdominal pain episodes.
* Recurrent dehydration with abdominal pain episodes requiring intravenous rehydration.
* Current personal diagnosis of depression or report of suicidality, mania or bipolar disorder.
* Family history of mania or bipolar disorder.
* Current use of opiates or other prescription pain medications and/or refusal to remain off opiate/prescription pain medications during the study period.
* Currently receiving additional therapies besides diet for recurrent abdominal pain and/or refusal to remain off such therapies during the study period, including but not limited to anticholinergic medications, antidepressant medications, biofeedback therapy, cognitive behavioral therapy.
* Hypersensitivity to SAM-e.
* Inability of child to provide assent and/or inability of parent/custodian to give consent.

Ages: 8 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2007-06; Primary Completion 2011-03 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeannie Huang, MD, MPH, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- SAM-e: This an open-labeled study. All participants received SAM-e.
  S-adenosyl methionine : All participants received oral SAM-e which was initiated at a dose of 200 mg daily and escalated by 200 mg every week to a maximum dose of 1400 mg daily if patients did not report significant resolution of abdominal pain (defined as reduction in reported pain and to a maximum frequency of once weekly).
Period: Overall Study
Arm/Group | SAM-e
Started | 8
Completed | 6
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- Sam-e (Treatment): This an open-labeled study. All participants will be part of the treatment group and receive SAM-e.
  S-adenosyl methionine : S-adenosyl methionine will be dosed as 200 mg tablets with doses ranging from 200 to 1400 mg daily.
Arm/Group | Sam-e (Treatment)
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Wong-Baker FACES Pain Rating Scale
Description: We scored the Wong-Baker Pain Rating Scale numerically on a scale of 0 (no pain) to 4 (worst pain).
Time Frame: 0, 2 weeks, 1 month, 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- SAM-e: This an open-labeled study. All participants will receive SAM-e.
  S-adenosyl methionine : S-adenosyl methionine will be dosed as 200 mg tablets with doses ranging from 200 to 1400 mg daily.
Arm/Group | SAM-e
Number analyzed (Participants) | 6
units on a scale
  Wong-Baker FACES Pain Rating Scale (2-months) | 3 (0)
  Wong-Baker FACES Pain Rating Scale (1-month) | 3 (0)
  Wong-Baker FACES Pain Rating Scale (2 weeks) | 4 (1)
  Wong-Baker FACES Pain Rating Scale (baseline) | 4 (0)
Statistical Analysis 1: Comparison: SAM-e; Test type: Non-Inferiority or Equivalence — No power calculation was calculated as this was a pilot study to determine such parameters; p = 0.004, MANOVA

2. Secondary Outcome: Safety
Description: Assessments of liver transaminases and alkaline phosphatasewere performed at baseline, 2 weeks, 1 month and 2 months. Depression and mania were assessed weekly.
Time Frame: 0, 2 weeks, 1 month, 2 month
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Sam-e (Treatment)
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 7/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sam-e (Treatment) (N=8)
headaches (Nervous system disorders) | 7
Alkaline Phosphatase Decrease (Hepatobiliary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No